CLINICAL TRIAL: NCT00126633
Title: A Study of Fixed-Dose Rate Gemcitabine, Cisplatin, and Bevacizumab in Previously Untreated Patients With Metastatic Pancreatic Cancer
Brief Title: Gemcitabine, Cisplatin, and Bevacizumab in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000437858; UCSF-04451; GENENTECH-AVF2937s
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: bevacizumab
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving gemcitabine and cisplatin together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine and cisplatin together with bevacizumab works in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine time to disease progression in patients with previously untreated metastatic adenocarcinoma of the pancreas treated with gemcitabine, cisplatin, and bevacizumab.
* Determine the safety and toxicity of this regimen in these patients.

Secondary

* Determine the objective response rate in patients treated with this regimen.
* Determine the efficacy of this regimen, in terms of the proportion of patients with ≥ a 50% decline in the CA19-9 biomarker, in these patients.
* Determine the median survival of patients treated with this regimen.
* Correlate serum markers of angiogenesis and circulating tumor micrometastases with clinical outcome of patients treated with this regimen.

OUTLINE: This is an open-label, non-randomized study.

Patients receive gemcitabine IV over 100 minutes, cisplatin IV over 30-60 minutes, and bevacizumab* IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients may receive additional study treatment at the discretion of the investigator.

NOTE: *Patients may continue to receive other components of therapy if bevacizumab is discontinued due to toxicity.

After completion of study treatment, patients are followed at 28 days and then monthly thereafter.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Must have documented extrapancreatic metastases

    * Radiographically measurable disease is not required
* Previously untreated disease
* No CNS or brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion or epoetin alfa [Epogen®] support allowed)
* No evidence of bleeding diathesis or coagulopathy

Hepatic

* INR ≤ 1.5 (except for patients receiving full-dose warfarin)
* Bilirubin ≤ 2.0 mg/dL
* AST or ALT ≤ 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)

Renal

* Creatinine ≤ 2.0 mg/dL
* Urine protein:creatinine ratio ≤ 1

Cardiovascular

* No New York Heart Association class II-IV congestive heart failure
* No myocardial infarction or stroke within the past 6 months
* No uncontrolled hypertension (i.e., blood pressure > 160/110 mm Hg despite antihypertensive therapy)
* No unstable angina
* No unstable symptomatic arrhythmia requiring medication

  * Patients with chronic atrial arrhythmia (i.e., atrial fibrillation or paroxysmal supraventricular tachycardia) are eligible
* No peripheral vascular disease ≥ grade 2

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No significant traumatic injury within the past 28 days
* No serious non-healing wound, ulcer, or bone fracture
* No other malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious systemic disease
* No history of any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that would preclude study treatment

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* More than 28 days since prior major surgery, or open biopsy
* More than 7 days since prior fine needle aspirations or core biopsies
* No concurrent major surgery

Other

* No prior therapy, including systemic or investigational therapy, for locally advanced or metastatic pancreatic cancer

  * Treatment given in the adjuvant setting (e.g., radiotherapy and/or chemotherapy, given either concurrently or systemically) is not considered prior therapy provided progressive disease occurred > 6 months after completion of prior treatment
* Concurrent continuation of therapeutic doses of warfarin or low-molecular weight heparin allowed for pulmonary embolism, deep vein thrombosis, atrial fibrillation, or other clinical indications provided patients has been on a stable dose for ≥ 28 days with no further clotting or bleeding complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-04; Primary Completion 2006-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Time to progression
Duration of response
Overall survival
Toxicity as measured by NCI CTC version 2.0
Micrometastases for predicting time to progression and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ko, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Result] Ko AH, Dito E, Schillinger B, Venook AP, Xu Z, Bergsland EK, Wong D, Scott J, Hwang J, Tempero MA. A phase II study evaluating bevacizumab in combination with fixed-dose rate gemcitabine and low-dose cisplatin for metastatic pancreatic cancer: is an anti-VEGF strategy still applicable? Invest New Drugs. 2008 Oct;26(5):463-71. doi: 10.1007/s10637-008-9127-2. Epub 2008 Apr 1. PMID 18379729